CLINICAL TRIAL: NCT03982095
Title: Survey on Lifestyle, Perceived Barriers and Development of Change in Patients With Prostate Cancer
Acronym: PCa_LS
Status: Completed | Type: Observational
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Collaborators: University of Modena and Reggio Emilia (Other)
Responsible Party: Sponsor
Other Study IDs: PCa_Oss_2019
Record Dates: First submitted 2019-05-08; First posted 2019-06-11 (Actual); Last update posted 2025-06-20 (Actual); Status verified 2021-11

CONDITIONS: Prostatic Neoplasm; Physical Activity; Health Behavior; Lifestyle, Sedentary
Keywords: Prostatic neoplasm; Physical therapy modalities; Healthy lifestyle; Biobehavioral Sciences
MeSH Terms: conditions — Prostatic Neoplasms; Motor Activity; Health Behavior; Sedentary Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Prostate cancer (PCa) is among the most widespread in the male population and represents 20% of all cancers diagnosed from the age of fifty, in Italy. Androgen deprivation therapy (ADT) is a common strategy of treatment that is used for increase survival. However, ADT is associated with significant side effects, such as fatigue, loss of muscle mass and strength, cognitive decline and reduced quality of life, with an increased the risk for falls and fractures, cardiometabolic syndrome and cardiovascular events.

The numerous side effects from ADT could potentially be countered by the regular Physical Exercise (PE), with favorable effects on body composition, physical performance, bone health and cognitive function.

However, to maintain the results obtained, PE must be undertaken regularly, becoming a healthy habit of life. The patient motivation is therefore a fundamental element for guaranteeing adherence to the intervention and its integration into people's lifestyle.

The study aim is to analyzed patients with PCa at the time of diagnosis regarding their lifestyle, includes regular PE, and motivation to make changes about their habits. In addition, the investigators will describe the perceived barriers by patients about this change.

The data collected will allow the development of an experimental intervention of PE, associated with therapeutic education, and assess its impact on the health of patient undergoing ADT, considering the realistic possibilities of application in the daily life of these patients, testing its feasibility and safety, the compliance and the satisfaction of the patients.

DETAILED DESCRIPTION:
Participants will be invited to an interview guided by open-ended questions, focused on collecting information related to the usual lifestyle, the motivation to undertake healthy changes and the perceived barriers to adopting an healthy lifestyle. In particular, the interview is focused on collecting the following information:

1. the level of PE: type, frequency and intensity;
2. the presence of health risk factors such as smoking, eating and drinking habits;
3. the presence of cognitive disorders, investigated through the Mini Mental State Examination and through some questions aimed at catching the subjective perception of one's cognitive state;
4. the stage of motivation to the adoption of healthy lifestyle that includes regular PE;
5. the perceived barriers to one's ability to change one's lifestyle by adopting a regular habit of PE.

During the interview, all patients will receive information about the importance of adopting a healthy lifestyle for the prevention of various diseases and even more to counteract the negative effects of PCa care. By adopting the Transtheoretical Model of Change (by Prochaska and DiClemente), will be identified the stage of motivation to change the risk factor identified through the interview. Consequently, these patients will receive a personalized message, with the aim of promoting change to healthy behavior. All patients will be informed about the existence and purpose of the Life Style Service in collaboration with LILT (Italian League for the Fight against Cancer) of the Health Information Service, active at CORE, at the Santa Maria Nuova Hospital in Reggio Emilia. In particular, patients in the "contemplation stage" will be informed about the possibility of contacting the clinic spontaneously at any time.The researcher will send the request to the public health clinic.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed with histologically documented prostate cancer;
* at least 18 years old;
* willing and able to give written informed consent;
* able to read and understand Italian Language;

Exclusion Criteria:

* patients undergoing major surgery in the three months prior to diagnosis of prostate cancer, which caused a change in lifestyle during the three months prior to PCa diagnosis

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible participants for this study are men with newly PCa diagnosis, possible candidates to radical prostatectomy, radiotherapy and/or androgen deprivation therapy. Patients will be enrolled from the community across the province of Reggio Emilia.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-09-04 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Identification the risk factor for health of the newly diagnosed patients with PCa | Baseline
  The presence of factors that influence healthy lifestyle will be identified throught a questionnaire with data and personal information, and clinical data: the stage of the tumor, ongoing/planned therapies, presence of comorbidity (Charlson index). The daily habits of patients, such as smooking, eating and drinking habits will be investigated with open question, with specific section about the level of PE performed (type, intensity and frequency).

SECONDARY OUTCOMES:
Investigation of the presence of cognitive disfunction | Baseline
  Date will be collected with the Mini Mental State Examination (MMSE) and through a questionnaire on the subjective perception of the prior cognitive state.
Investigation the motivation to change and perceived barriers | Baseline
  The influence of risk factor for health status, the motivation to change and the perceived barriers will be identified with a specific guided interview by the Prochaska and DiClemente's Transtheoretical Model (Stages of Change).

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Costantini, Dr, Study Chair — Azienda Unità sanitaria Locale - IRCCS di Reggio Emilia
Locations (1):
- Azienda USL - IRCCS, Reggio Emilia, Italy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bressi B, Iotti C, Cagliari M, Fugazzaro S, Cavuto S, Bergamaschi FAM, Moscato A, Costi S. Physical exercise habits, lifestyle behaviors, and motivation to change among men with prostate cancer: a cross-sectional study. Support Care Cancer. 2022 Jun;30(6):5017-5026. doi: 10.1007/s00520-022-06911-z. Epub 2022 Feb 22. PMID 35194723